CLINICAL TRIAL: NCT07345104
Title: Accuracy of Digital Mandibular Repositioning in Occlusal Reconstruction for Patients With Disc Displacement: A Randomized Controlled Trial
Brief Title: Accuracy of Digital Mandibular Repositioning in Occlusal Reconstruction for Patients With Disc Displacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Associate Professor & Associate Dean, Dept. of Prosthodontics, Fujian Medical University; Adjunct Associate Professor, Dept. of Applied Prosthodontics, Nagasaki University, Nagasaki, Japan., Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024GGA070
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Disc Displacement
Keywords: Reducible disc displacement; Mandibular repositioning; Occlusal splint therapy; Digital dentistry; CBCT; Electronic facebow

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of four parallel groups based on patient preference and clinical feasibility (non-randomized allocation):
  * Group A (Intraoral Direct Positioning): Therapeutic mandibular position determined by clinical clicking elimination method.
  * Group B (Articulator Positioning): Therapeutic position determined using semi-adjustable articulator with facebow transfer and condylar guidance records.
  * Group C (Digital Anatomical Positioning): Therapeutic position determined by integrating intraoral scanning, CBCT, and MRI data using CAD software.
  * Group D (Digital Jaw Motion Tracking): Therapeutic position determined
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding and Masking Procedures:
  1. Outcome Assessor Blinding
     * All clinical and radiographic outcome measurements will be performed by independent assessors who are unaware of the participant's group allocation.
     * Participants will be assigned unique, randomly generated identification codes that do not reveal group assignment.
     * Radiographic images (CBCT and MRI) will be anonymized and presented in a randomized order to blinded radiologists.
  2. Limitations of Masking
     o Complete blinding is not possible due to the distinct nature of interventional approaches: a) Participants will be aware of their specific mandibular repositioning technique b) Clinicians performing interventions cannot be blinded due to different positioning methods
  3. Blinding Process for Outcome Assessment o Clinical outcome measures (Craniomandibular Index, Joint Movement Assessment) will be evaluated by a research assistant not involved in the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intraoral Direct Positioning (Active Comparator): Therapeutic mandibular position is determined using the clinical clicking elimination method. Patients perform wide opening until clicking occurs, then gradually retract the mandible while making opening-closing movements to identify the minimal protrusion position without clicking. A repositioning splint is fabricated based on this position.
  Interventions: Device: Clinical Clicking Elimination Repositioning Splint
- Articulator Positioning (Experimental): Therapeutic mandibular position is determined using a semi-adjustable articulator (Artex CR) with mechanical facebow transfer. Condylar guidance angles are obtained from protrusive and lateral excursion records. The optimal position is calculated based on CBCT joint space measurements and MRI disc displacement data. A repositioning splint is fabricated accordingly.
  Interventions: Device: Adjustable Articulator Repositioning Splint
- Digital Anatomical Positioning (Experimental): Therapeutic mandibular position is determined by integrating intraoral scanning data with CBCT-reconstructed 3D jaw models using CAD software (Exocad). The optimal position is calculated by referencing MRI disc reduction phase, ideal joint space ratios (anterior:superior:posterior = 1:1.3:1), and anatomical landmarks. A repositioning splint is digitally designed and 3D-printed.
  Interventions: Device: CAD-Designed Anatomical Repositioning Splint
- Digital Jaw Motion Tracking (Experimental): Therapeutic mandibular position is determined by integrating 3D jaw models with electronic jaw tracking data (Zebris JMA system). The optimal position is identified by analyzing condylar movement trajectories, specifically locating the crossover points of the "figure-8" pattern indicating disc displacement, combined with dynamic MRI and joint space parameters. A repositioning splint is digitally designed and 3D-printed.
  Interventions: Device: Electronic Jaw Tracking Repositioning Splint

INTERVENTIONS:
Device: Clinical Clicking Elimination Repositioning Splint — A custom-fabricated hard acrylic repositioning splint based on manual intraoral mandibular positioning. The splint is created by:
  1. Clinically identifying the optimal jaw position through clicking elimination technique
  2. Taking alginate impressions of maxillary and mandibular arches
  3. Pouring stone models and manually adjusting mandibular model to the determined position
  4. Fabricating a hard acrylic splint with 1-2 mm occlusal clearance
  5. Finishing and polishing the splint Patients wear the splint 24 hours daily (except during meals) for 3 months, with adjustments at 2 weeks, 1 month, 2 months, and 3 months.
  Arms: Intraoral Direct Positioning
Device: Adjustable Articulator Repositioning Splint — A custom-fabricated hard acrylic repositioning splint using adjustable articulator (Artex CR) methodology:
  1. Performing mechanical facebow transfer
  2. Recording condylar guidance parameters in protrusive and lateral excursions
  3. Analyzing CBCT joint space measurements and MRI disc displacement data
  4. Mounting study models on Artex CR articulator with precise condylar settings
  5. Manually adjusting splint to achieve optimal mandibular position
  6. Fabricating hard acrylic splint with 1-2 mm occlusal clearance Patients wear the splint 24 hours daily (except during meals) for 3 months, with adjustments at 2 weeks, 1 month, 2 months, and 3 months.
  Arms: Articulator Positioning
Device: CAD-Designed Anatomical Repositioning Splint — A digitally designed and 3D-printed repositioning splint using advanced digital workflow:
  1. Performing intraoral digital scanning (iTero Element)
  2. Acquiring CBCT scan (I-CAT FLX)
  3. Importing MRI disc displacement data
  4. Using CAD software (Exocad) to:
     * Overlay intraoral scan with CBCT 3D model
     * Reference MRI disc reduction phase
     * Calculate optimal joint space ratios
  5. Digitally designing splint with precise mandibular positioning
  6. Fabricating hard acrylic splint with 1-2 mm occlusal clearance Patients wear the splint 24 hours daily (except during meals) for 3 months, with adjustments at 2 weeks, 1 month, 2 months, and 3 months.
  Arms: Digital Anatomical Positioning
Device: Electronic Jaw Tracking Repositioning Splint — A digitally designed repositioning splint using electronic jaw motion tracking:
  1. Performing 3D jaw motion tracking (Zebris JMA system)
  2. Capturing mandibular movement trajectories
  3. Identifying "figure-8" pattern crossover points indicating disc displacement
  4. Integrating dynamic MRI data
  5. Analyzing optimal joint space parameters
  6. Using CAD software to design precise mandibular positioning splint
  7. Fabricating hard acrylic splint with 1-2 mm occlusal clearance Patients wear the splint 24 hours daily (except during meals) for 3 months, with adjustments at 2 weeks, 1 month, 2 months, and 3 months.
  Arms: Digital Jaw Motion Tracking

SUMMARY:
This study evaluates a new, individualized treatment for adolescents with temporomandibular joint disorders (TMD) caused by bilateral, reducible disc displacement. Participants will undergo clinical and imaging examinations, including cone-beam CT (CBCT), MRI, and intraoral digital scanning to create three-dimensional models of the teeth and jaw. Based on these data, the study team will design and fabricate a personalized repositioning digital occlusal splint for each participant. Patients will be instructed on how to wear the splint and will return for regular follow-up visits to monitor symptoms and adjust the splint as needed. The study aims to improve pain, chewing function, and overall quality of life. All research-related imaging, digital scans, splint fabrication, and follow-up visits will be provided at no cost to participants. Possible risks include temporary discomfort or pressure when first wearing the splint, and the possibility that symptoms may not improve as expected. Participant safety, privacy, and data confidentiality will be strictly protected, and participants may withdraw from the study at any time without affecting their future medical care.

DETAILED DESCRIPTION:
Detailed Description This study evaluates four different methods for mandibular repositioning in patients with bilateral reducible temporomandibular joint (TMJ) disc displacement requiring occlusal reconstruction.

Methods of Mandibular Repositioning:

1. Intraoral Direct Positioning Group: The therapeutic jaw position is determined clinically using the clicking elimination method, where patients open wide until clicking occurs, then gradually retract the mandible while performing opening-closing movements to find the minimal protrusion position without clicking.
2. Articulator Positioning Group: Uses mechanical facebow transfer and semi-adjustable articulator (Artex CR) with condylar guidance parameters obtained from protrusive and lateral excursion records. The therapeutic position is determined by analyzing CBCT joint space measurements and MRI disc displacement data.
3. Digital Anatomical Positioning Group: Combines intraoral scanning data with CBCT-reconstructed 3D jaw models. The therapeutic position is determined by referencing MRI disc reduction phase, optimal joint space ratios, and anatomical landmarks using CAD software (Exocad).
4. Digital Jaw Motion Tracking Group: Integrates 3D jaw models with electronic jaw tracking data (Zebris). The therapeutic position is determined by analyzing condylar movement trajectories (identifying the "figure-8" pattern crossover points indicating disc displacement) combined with dynamic MRI and optimal joint space parameters.

Treatment Protocol: All groups receive digitally designed and manufactured repositioning splints. Patients wear splints 24 hours daily (except during meals) for 3 months, with follow-up adjustments at 2 weeks, 1 month, 2 months, and 3 months.

Imaging Protocol:

* CBCT (I-CAT FLX): 120 kV, 5 mA, 0.2 mm resolution
* MRI (GE Discovery MR750w 3.0T): Bilateral TMJ surface coils, oblique sagittal and coronal views in closed-mouth position, oblique sagittal in maximum opening

Assessment Methods:

* Joint space measurements using Ikeda's method on registered pre- and post-treatment CBCT images
* Condyle position analysis using Gelb 4/7 position criteria
* Disc-condyle angle measurement on MRI (>15° defined as disc displacement)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of reducible temporomandibular joint (TMJ) disc displacement according to the 2014 revised criteria of the International Association for Dental Research;
2. Bilateral reducible disc displacement confirmed by MRI;
3. Reproducible joint clicking during mandibular opening and closing;
4. Permanent dentition with full cognitive and communicative ability;
5. Signed informed consent with good treatment compliance.

Exclusion Criteria:

1. Non-reducible disc displacement, osteoarthrosis, isolated myofascial pain, or other conditions not meeting diagnostic criteria;
2. Receipt of other TMJ disorder treatments within the past 3 months;
3. Presence of systemic diseases, psychiatric disorders, or impaired consciousness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Temporomandibular Joint Space Ratio | Baseline and 3 months post-treatment
  Quantitative assessment of changes in temporomandibular joint space using Cone Beam Computed Tomography (CBCT) with Ikeda's method.
Change in Disc-Condyle Relationship Angle | Baseline and 3 months post-treatment
  Quantitative assessment of disc displacement using Magnetic Resonance Imaging (MRI) with angle measurement technique.

CONTACTS AND LOCATIONS:
Locations (1):
- School and Hospital of Stomatology, Fujian Medical University,, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No